CLINICAL TRIAL: NCT01472068
Title: A Pilot Study to Evaluate the Safety and Performance of Neuromuscular Electrical Stimulation (NMES) With the Inko RS Device for the Treatment of Stress Urinary Incontinence
Brief Title: A Pilot Study to Evaluate Safety and Performance of Neuromuscular Electrical Stimulation With the Inko RS Device for the Treatment of Stress Urinary Incontinence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Medical Research, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMR-11-1014
Record Dates: First submitted 2011-11-09; First posted 2011-11-16 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Stress Urinary Incontinence
Keywords: Incontinence; NMES
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inko RS device (Experimental): 30 minutes of treatment with the Inko RS device, five days each week, for 12 weeks.
  Interventions: Device: Inko RS Device

INTERVENTIONS:
Device: Inko RS Device — 30 minute pre-programmed treatment for 5 days out of 7. Treatment to be carried out while standing.

SUMMARY:
This is a pilot clinical study taking place at one site in Berlin, Germany using Neuromuscular Electrical Stimulation (NMES) to stimulate the pelvic floor muscles of 20 women suffering from stress urinary incontinence. This involves a 12 week, 30 minute, 5 days out of 7 set treatment program with the device. After the 12 week treatment programme the subjects will be asked to perform daily set exercises for a further 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are female and at least 18 years of age.
* Subject has signed informed consent form prior to any study related activity
* Subjects who have previously failed a 6 week volitional pelvic floor muscle training program.
* Subjects who have been clinically diagnosed with stress urinary incontinence and demonstrate a >4g urine leakage following a standardised 1-minute stress test at 1 hour post-bladder filling protocol (1-hour pad weight test). Stress urinary incontinence is defined as complaint of involuntary leakage on effort or exertion, or on sneezing and coughing' (International Continence Society).
* Subjects who have scored at least 18 out of 27 for the Stress Incontinence Questions and are confirmed as having predominant stress urinary incontinence on the Medical, Epidemiologic and Social Aspects of Aging Urinary Incontinence (MESA) Questionnaire completed at the screening assessment.
* Subjects with a Body Mass Index of < 30 kg/m2
* Subjects who are able to give voluntary, written informed consent to participate in this study and from whom consent has been obtained.
* Subjects who are able to understand this study and are willing to complete all the study assessments.

Exclusion Criteria:

* Subjects who have an existing medical condition that would compromise their participation in the study.
* Subjects who have a physical condition that would make them unable to perform the study procedures.
* Subjects who have or a history of any respiratory condition including a chronic cough.
* Subjects with a history of an underlying neurological condition.
* Subjects with a history of low back pain involving the spinal nerve root.
* Subject who are currently taking medication, or have taken medication in the last 4 weeks, for urinary incontinence or that effect urinary output function including anti-cholinergics or anti-histamines or any anti-anxiety medications.
* Subjects with a blood clotting disorder or who are taking anti-coagulant medications.
* Subjects who have previously had any uro-gynaecological related surgery excluding hysterectomy.
* Subjects with a clinical diagnosis of prolapse greater than Stage 2.
* Subjects who are pregnant or could be pregnant.
* Subjects who are less than 6 months post-partum or who are lactating.
* Subjects who have any intra-uterine devices or metal implants in the pelvic area, including hip and lumbar spine.
* Subjects with pelvic pain or fibromyalgia or paravaginal defect.
* Subjects with an active implanted medical device (ie pacemaker, pump etc).
* Subjects with a history of heart disease or stroke.
* Subjects with a known cancer.
* Subjects with an injury or disability affecting any part of their body which will be in contact with the garment.
* Subjects who are currently involved in any injury litigation claims.
* Subjects who have participated in a clinical study in the last 3 months.
* Any vulnerable subjects defined as individuals whose willingness to volunteer in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate. Examples are members of a group with a hierarchical structure, such as medical, pharmacy, dental, and nursing students, subordinate hospital and laboratory personnel, employees of the pharmaceutical and medical device industry, members of the armed forces, and persons kept in detention. Other vulnerable subjects include patients with incurable diseases, persons in nursing homes, unemployed or impoverished persons, patients in emergency situations, ethnic minority groups, homeless persons, nomads, refugees, minors, and those incapable of giving consent.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Based on a reduction in urine leakage following a standardised 1- min stress test at 1 hour post-bladder filing protocol (1-hour pad weight test) at 12 weeks compared to baseline following a 12 week treatment programme with the Inko RS Device. | 12 weeks

SECONDARY OUTCOMES:
To evaluate an improvement in quality of life assessed using the Incontinence Quality of Life Questionnaire (I-QOL). | 4 wks, 8 wks and 12 weeks
Evaluate an improvement in quality of life assessed using the Medical, Epidemiologic and Social Aspects of Aging Urinary Incontinence Questionnaire (MESA) | at 4, 8 and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- St. Hedwig Krankenhaus, Berlin, State of Berlin, Germany